CLINICAL TRIAL: NCT03312062
Title: Influence of Foam Rolling on Elbow Proprioception, Strength, and Functional Motor Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Fatma Özden, PT, Physical Therapist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3399-GOA
Record Dates: First submitted 2017-09-28; First posted 2017-10-17 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Proprioceptive Disorders
Keywords: elbow; foam rolling; proprioception; motor performance; strength
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: There are 2 groups. Study group will receive foam rolling exercise. Control group will receive no foam rolling exercise. They will be handed a brochure about the proprioception and its role in injury prevention and foam rolling . Study group will be evaluated before foam rolling exercise . Afterwards, second evaluation will be performed after 4 weeks and follow up after 4 more weeks. Control group will be evaluated for the first time. Afterwards, second evaluation will be performed after 4 weeks and follow up after 4 more weeks.
Who Masked: Participant
Masking Description: All of participants must be healthy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam Rolling Group (Experimental): The participants in this group will receive foam rolling exercise.
  Interventions: Other: Foam Rolling Exercise
- Control Group (No Intervention): The participants in this group will receive no foam rolling. They will only be evaluated.

INTERVENTIONS:
Other: Foam Rolling Exercise — Foam rolling exercise will be performed actively. Participants will use a foam roller for exercise. They will position the foam roller on the chair. Afterwards, they will use their body weights to rub the elbow area (biceps brachii muscle) with this foam. There will be 2 sets and each set will be 1 minute. Single set contains 10 repetitions in 1 minute with 30 seconds resting period between sets.
  Arms: Foam Rolling Group

SUMMARY:
The purpose of this study is to investigate the long-term effects of foam rolling on elbow proprioception, strength and functional motor performance with healthy participants . Study group will receive foam rolling exercise. Control group will receive no foam rolling exercise. Control group will be given a brochure including information about proprioception and foam rolling.

DETAILED DESCRIPTION:
There is no information in literature about the effects of foam rolling on elbow proprioception, strength and functional motor performance. The purpose of this study is to investigate long-term effects of foam rolling with healthy participants. Study group will receive foam rolling exercise actively by themselves on elbow.

Foam rolling exercise will be applied 10 times each for 1 minute. These exercises will be performed as 2 sets. After each set will be a resting period for 30 seconds.A total of 12 sessions of exercise will be performed three times a week. Second evaluation will be performed after 4 weeks. Then the follow up evaluation (third evaluation) will be performed 4 weeks later. Control group will receive no foam rolling exercise. They will be handed a brochure about the proprioception and its role in injury prevention and foam rolling. Control group will be evaluated for the first time. Afterwards, second evaluation will be performed after 4 weeks and follow up after 4 more weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above healthy participants
* No pain in elbow area within 6 months and at the time of measurement
* To be able to complete all evaluations and applications to be carried out

Exclusion Criteria:

* Having previous foam rolling and self-myofascial relaxation applications on the target area
* Having acne and similar skin problems, open wounds
* Having upper extremity injury, history of fracture or surgery
* Having any systemic musculoskeletal disease
* Having diagnosis of diabetic mellitus or peripheral neuropathy
* Having osteoporosis diagnosis
* Having any cardiovascular disease
* Having vertigo
* Being pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Elbow Proprioception | Baseline, after 4 weeks foam rolling exercise period and then follow up measurement 1 month
  Change of elbow joint position sense (with digital inclinometer in degree) and force match ( hand held dynamometer in kg )

SECONDARY OUTCOMES:
Biceps Brachii Strength | Baseline, after 4 weeks foam rolling exercise period and then follow up measurement 1 month
  Change of biceps brachii strength ( hand held dynamometer in kg )
Elbow Functional Motor Performance | Baseline, after 4 weeks foam rolling exercise period and then follow up measurement 1 month
  Change of elbow functional motor performance (push up test, modified pull up test, closed kinetic chain upper extremity stability test )

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, Study Director — Dokuz Eylul University
Locations (1):
- Fatma Özden, Izmir, Bornova, Turkey (Türkiye)